CLINICAL TRIAL: NCT00153907
Title: A Phase I Study of Oral Navelbine and Capecitabine in the Treatment of Metastatic Breast Cancer
Brief Title: Navelbine and Capecitabine in the Treatment of Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Craig A. Bunnell, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-217
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Xeloda; Navelbine; capecitabine; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

INTERVENTIONS:
Drug: Navelbine — Given orally on day 1 and 8 of each cycle, dose will vary. If participant is at highest dose they will take navelbine on day 1, 8 and 15 until disease progression or unacceptable side effects occur.
Drug: Capecitabine — Taken twice a day on days 1-14 until disease progression or unacceptable side effects occur.
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to find the highest dose of capecitabine and oral navelbine that can be given without causing severe side effects, and to determine the safety, tolerability, and effects (good and bad) of capecitabine given with oral navelbine to patients with advanced breast cancer.

DETAILED DESCRIPTION:
* Not every patient will be receiving the same dose of capecitabine and navelbine. A small group will be enrolled onto the study and given certain doses of each drug. If they tolerate them well (have few or easily manageable side effects), the next small group of people enrolled will receive a higher dose of one of the drugs. This will continue until we find the highest doses of the drugs that can be given without causing serious or unmanageable side effects.
* Patients will be given oral navelbine on days 1 and 8 of each cycle, unless they are at the highest dose. In which case, they will be given navelbine on days 1, 8 and 15. Capecitabine will be given on days 1-14 of each cycle in two divided doses approximately 12 hours apart.
* While patients are on the study they will have the following tests and procedures performed: physical examination every 3 weeks; routine blood work every week; extensive laboratory tests every 3 weeks; disease status will be checked every 6 weeks (2 cycles) unless there are symptoms of disease progression.
* The weekly treatment will continue unless there is disease progression or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer with evidence of locally advanced or metastatic disease
* Female patients age 18 or older
* No more than three prior chemotherapeutic regimens in the metastatic setting
* ANC > 1,500/mm3
* Platelet count > 100,000/mm3
* SGOT < 3 x ULN
* Bilirubin < 1.5 x ULN
* Performance status of 0 or 1
* At least 3 weeks since prior chemotherapy or 2 weeks since prior radiation, surgery or any anticancer investigational agent
* Able to swallow and retain oral medications
* Measurable disease

Exclusion Criteria:

* Prior vinca alkaloids
* Active gastrointestinal disease or disorder
* Pregnant or lactating
* Serious co-morbid medical or psychological condition
* Prior bone marrow or stem cell transplant
* Prior documented severe sensitivity to 5-FU

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To define the maximally tolerated dose and evaluate the feasibility and toxicity of capecitabine and oral navelbine administered in combination. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Bunnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts